CLINICAL TRIAL: NCT05739968
Title: Impacts and Testing of the "Multi-domains Active-living Program (MAP)" in Newly Diagnosed Operable Non-Muscle Invasive Bladder Cancer Patients - Current Status and the Effects of Combining With eHealth-Enhanced Randomized Controlled Trial
Brief Title: Impacts and Testing of the "Multi-domains Active-living Program" in Operable Non-Muscle Invasive Bladder Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 201912156RIND
Record Dates: First submitted 2023-01-26; First posted 2023-02-22 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Bladder Cancer; Quality of Life
Keywords: Bladder Cancer; Personalized Supportive Cancer Care Program; Physical symptom; Fear of cancer recurrence; Physical function; Sexual/intimacy; Physical activity
MeSH Terms: conditions — Urinary Bladder Neoplasms; Coitus; Motor Activity | interventions — oncomodulin

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled clinical trial which to compare the effects of the OCM care only (control) vs. MAP+OCM program (experimental group) on non-muscle invasive bladder cancer (NMIBC) patients.
  For both groups, we assessed patients' outcomes (including baseline data) for 5 times (T1=baseline/during hospitalization of receiving surgery & before their hospital; T2 to T5 = 6±2 weeks, 3, 6, 12 months after operation).
Who Masked: Participant, Care Provider, Investigator
Masking Description: This study was not fully blinded; however, the group allocation was concealed from the patient and primary researcher until after baseline assessments were completed. A primary researcher obtained patient consent, collected self-reported assessments, and if the patients were randomized to intervention group, the intervention trainer explained the MAP program to participants. The study statistician and data managers remained blinded at all times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Control Group: Usual care + oncology case manager (OCM) care, UC group or Control group
  Interventions: Other: Usual care + oncology case manager (OCM) care
- experimental group (Experimental): The experimental group is Multi-domains Active-living Program (MAP) with e-health enhanced intervention + usual care + oncology case manager (OCM) care. Main contents of MAP are to (a) cope multi-domain of distress, and (b) develop an active life style to handle their life after cancer, including effective coping, relaxation, regular physical activities, and balance nutrition. Four face-to face interventions will be delivered, including: day before hospital discharge post-operation, before the last weekly instillations of induction therapy (around 6±2 weeks post operation), 2nd-time cystoscopy and before 1st maintenance therapy (around 3- month post operation) and 3rd-time cystoscopy which before the second cycle of maintenance therapy (around 6- month post operation) [section 1-4], respectively.
  Interventions: Other: Multi-domains Active-living Program (MAP) with e-health enhanced intervention + usual care + oncology case manager (OCM) care

INTERVENTIONS:
Other: Usual care + oncology case manager (OCM) care — Usual care + oncology case manager (OCM) care
  Arms: control group
Other: Multi-domains Active-living Program (MAP) with e-health enhanced intervention + usual care + oncology case manager (OCM) care — Multi-domains Active-living Program (MAP) with e-health enhanced intervention + usual care + oncology case manager (OCM) care
  Arms: experimental group

SUMMARY:
Among bladder cancer, the majority of them (70%) are non-muscle-invasive bladder cancer (NMIBC). The survival time is even longer in NMIBC. Patients with NMIBC receive surgery or transurethral resection of bladder tumor (TURBT). However, patients with NMIBC need to receive a three-month repeatedly intrusive cystoscope from diagnosis for the first year. Furthermore, following each cystoscope, patients will receive 3 to 6 times bladder BCG (Bacille Calmette Guérin) or chemotherapy. These repeatedly intrusive cystoscopes, TURBT, and intensive bladder treatments might cause impacts on patients' life. The investigator aims to (1) construct a Multi-domains Active-living Program (MAP) with e-health enhanced intervention; and (2) compare the effects of the MAP with oncology case manager (OCM) care (experimental group) and OCM care only (control group) on the indicators and quality of life.

Intervention study is a 12-month two-group randomized trial, including OCM care only (control), Vs. MAP+OCM program (experimental group). MAP will be constructed based on literature review and preliminary results. Main contents of MAP are to (a) cope multi-domain of distress, and (b) develop an active life style to handle their life after cancer, including effective coping, relaxation, regular physical activities, and balance nutrition. Four face-to face interventions will be delivered, including: day before hospital discharge post-operation, before the last weekly instillations of induction therapy (around 6±2 weeks post operation), 2nd-time cystoscopy and before 1st maintenance therapy (around 3- month post operation) and 3rd-time cystoscopy which before the second cycle of maintenance therapy (around 6- month post operation) [section 1-4], respectively. A brief and automatic app reminder (before) and side-effect follow-up (after) from 2nd section of face-to face intervention will be sent. Boosting health education will also be provided by app/ phone calls or in person around 2 to 4 weeks after discharge. Patients in the MAP+OCM group also can raise their questions through APP to receive brief intervention. The outcomes will be assessed at 5 time points: time before first intervention, before 2nd to 4th interventions, and 12 months, T1-T5, respectively. We will use Generalized Estimated Equation (GEE) to analyze the data with total 120 subjects (60 Vs 60 estimated).

DETAILED DESCRIPTION:
Background: Non-muscle invasive bladder cancer (NMIBC) covers the majority of bladder cancer incidence. Operable NMIBC patients have to receive Transurethral Resection of Bladder Tumor (TURBT), every-three-month repeated cystoscopes and bladder-irrigated chemotherapy in the first year. The intrusion, repeated cystoscope/treatments and recurrence concern may influence NMIBC patients' quality of life.

Purposes: This is a 2-phase study. The aim of Phase I (first year) is to (1) test the psychometrics of NMIBC-specific Quality of Life (QOL) questionnaire "EORTC QLQ NMIBC 24-Chinese"; (2) examine patients' distress across multi-domains, including impacts on QOL, symptoms, physical function (upper/lower leg muscle power, balance), sexual/intimacy, fear of recurrence, and physical activity. Phase II (2nd&3rd year) is a two-group randomized trial for newly diagnosed NMIBC patients. It aims to (1) construct a Multi-domains Active-living Program (MAP) with e-health enhanced intervention; and (2) compare the effects of the MAP with oncology case manager (OCM) care (experimental group) and OCM care only (control group) of the effects on the above indicators (phase I) and the number of unexpected hospital visits.

Methods: Phase I is an instrument validation study. The "EORTC QLQ-NMIBC24-Chinese" will be to develop and examine of its psychometrics. We will also explore the above mentioned domains of QOL, distress, care needs, frequency of taking physical activities, etc. by questionnaire interview/assessment; and objective physical function measures (low leg muscle strengths and balance ability). An estimated sample size is 240 subjects. Phase II is a 12-month two-group randomized trial, including OCM care only (control), Vs. MAP+OCM program (experimental group). MAP will be constructed based on literature review and preliminary results. Main contents of MAP are to (a) cope multi-domain of distress, and (b) develop an active life style to handle their life after cancer, including effective coping, relaxation, regular physical activities, and balance nutrition. Four face-to face interventions will be delivered, including: day before hospital discharge post-operation, before the last weekly instillations of induction therapy (around 6±2 weeks post operation), 2nd-time cystoscopy and before 1st maintenance therapy (around 3- month post operation) and 3rd-time cystoscopy which before the second cycle of maintenance therapy (around 6- month post operation) [section 1-4], respectively. A brief and automatic app reminder (before) and side-effect follow-up (after) from 2nd section of face-to face intervention will be sent. Boosting health education will also be provided by app/ phone calls or in person around 2 to 4 weeks after discharge. Patients in the MAP+OCM group also can raise their questions through APP to receive brief intervention. The outcomes will be assessed at 5 time points: time before first intervention, before 2nd to 4th interventions, and 12 months, T1-T5, respectively. We will use Generalized Estimated Equation (GEE) to analyze the data with total 120 subjects (60 Vs 60 estimated).

Expected Outcome: This is the first study to test EORTC QLQ-NMIBC24 Chinese version, patients' distress and physical function as well as construct and test of a multi-domain MAP program. It would help us further build up evidence-based care and generalize to bladder cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* age ≥20 years
* operable newly diagnosed NMIBC patients who know their diagnosis and do not receive cystectomy (still keep their own bladder)
* patients can verbally communicate with others
* Mandarin / Chinese-reading and speaking

Exclusion Criteria:

* patients who has inoperable bladder cancer
* patient who has muscle invasive bladder cancer (MIBC) with expected cystectomy surgery in the time of diagnosed
* primary cancer unknown
* conscious unclear

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Quality of Life (consisting of symptoms, function, and health status) | The outcomes will be assessed at 5 time points: day before hospital discharge post-operation(Day 0), around 6±2 weeks post operation, around 3-month, 6-month and 12-month post operation.
  Quality of life will be assessed by the EORTC-QLQ. This Instrument is consists of 30 items to measure three subscales, includes 2 items global health status/quality of life, 15 items functional domains and 13 items cancer common related symptoms or problems. Two items in global health status use a 7-point summated scale (1 = poor; 7 = excellent) and other items are rated on 4-point Likert's Scales (1=not at all; 4=very much). The scores will be transformed to a range from 0 to 100. In global health status and functional domains, the higher scores indicate better function. In the symptoms subscale, lower scores indicate less severe symptoms (Aaronson et al., 1993). The Taiwan Chinese version has been demonstrated to be both reliable and valid (Chie et al., 2004).
Changes in Anxiety | The outcomes will be assessed at 5 time points: day before hospital discharge post-operation(Day 0), around 6±2 weeks post operation, around 3-month, 6-month and 12-month post operation.
  The severity of NMIBC patients' anxiety will be measured by the self-reporting Generalized Anxiety Disorder-7 (GAD-7).
  GAD is developed by Spitzer et al. (2006) and was used in a large primary care patient sample (Kroenke et al., 2007; Remes et al., 2016). The GAD-7 is a 7-item anxiety scale and is specifically linked to the DSM-IV (Text Revision) criteria (Spitzer et al., 2006). Response options were "not at all (score=0)," "several days (score=1)," "more than half the days (score=2)," and "nearly every day (score=3)," and the total GAD-7 score range is 0 to 21. The GAD-7 has good internal consistency (Cronbach α = 0.92) and test-retest reliability (intraclass correlation = 0.83) (Spitzer et al., 2006).
Changes in Depression | The outcomes will be assessed at 5 time points: day before hospital discharge post-operation(Day 0), around 6±2 weeks post operation, around 3-month, 6-month and 12-month post operation.
  The severity of NMIBC patients' depression will be measured by the self-reporting Patient Health Questionnaire-9 (PHQ-9).
  PHQ-9 is form a three page the Patient Health Questionnaire (PHQ) and is the 9-item depression module from the full PHQ (Kroenke et al., 2001). This questionnaire is used to screen for depression in primary care and other medical settings and with good sensitivity and specificity (Levis et al., 2019). In each PHQ-9 component, the lowest score is 0 (not at all), the highest score is 3 (nearly every day) and the total PHQ score range is 0 to 27.
Changes in Fear of Cancer Recurrence | The outcomes will be assessed at 5 time points: day before hospital discharge post-operation(Day 0), around 6±2 weeks post operation, around 3-month, 6-month and 12-month post operation.
  The 7-item Fear of Cancer Recurrence (FCR7) is a unidimensional instrument to assess cancer patients' concern regarding the coming back or progression of cancer. The FCR7 comprises 4 items measuring the severity of worry about recurrence, 2 items measuring the interference caused by FCR, and 1 item assessing the patient's response to FCR. The first 6 items are scored from 1 (not at all) to 5 (all the time) with higher scores indicating higher levels of FCR. The last item assessing the interference of FCR is scored from 1 (not at all) to 10 (a great deal) with the higher the score, the more the interference. The Chinese version of FCR7 has been validated and proven reliable with overall Cronbach's alpha being 0.90 (Lee et al., 2019).
Changes in Sleep Quality (consisting of sleep duration, sleep disturbances, sleep latency, daytime functioning, habitual sleep efficiency, subjective sleep quality, and sleep medication) | The outcomes will be assessed at 5 time points: day before hospital discharge post-operation(Day 0), around 6±2 weeks post operation, around 3-month, 6-month and 12-month post operation.
  The PSQI, which was developed by Buysee in 1989, is used to assess sleep quality on participants' sleep experiences during the past week (Buysse, Reynolds, Monk, Berman, & Kupfer, 1989). The PSQI is included seven component scores which are sleep duration, sleep disturbances, sleep latency, daytime functioning, habitual sleep efficiency, subjective sleep quality, and sleep medication. In each PSQI component, the lowest score is 0 (better), and the highest score is 3 (worse). The total PSQI score range is from 0 to 21, and the higher the score the worse the sleep. If the total PSQI score is more than 5, the result means the person has sleep problems (Buysse et al.,1989; He et al., 2015;Van Onselen et al., 2010). Both the original as well as the Chinese version of the Pittsburgh Sleep Quality Index (CPSQI) have good reliability and validity. In CPSQI, Cronbach's a coefficient for the hospital sample and test-retest reliability were 0.83 and 0.85, respectively (Tsai et al., 2005).
Changes in Physical Activity | The outcomes will be assessed at 5 time points: day before hospital discharge post-operation(Day 0), around 6±2 weeks post operation, around 3-month, 6-month and 12-month post operation.
  The Godin Leisure-Time Exercise Questionnaire (GLTEQ) is a simple tool to measure and classify cancer patients' levels of physical activity. The GLTEQ assesses types of leisure-time PA (LTPA) and their frequency and intensity over the previous 7 days. A total GLTEQ score is calculated as: (frequency of mild exercise×3) + (frequency of moderate exercise×5) + (frequency of strenuous exercise×9) (Godin, 2011; Godin & Shephard, 1985). The GLTEQ score has been proven to have the optimum discriminant functions in classifying percentile of body fat and percentile of maximum oxygen intake (Godin & Shephard, 1985).
Changes in Nutrition Status | The outcomes will be assessed at 5 time points: day before hospital discharge post-operation(Day 0), around 6±2 weeks post operation, around 3-month, 6-month and 12-month post operation.
  Mini Nutritional Assessment (MNA) is a comprehensive nutritional assessment scale for the past three months, including anthropometry (body mass index, brachial circumference, calf circumference, skinfold width of the triceps and subscapular muscles), dietary intake, functional geriatric assessment (mini-mental state examination, activities of daily living). The questionnaire includes 18 items with a total score of 0-30 points. The sum of the MNA score distinguishes between elderly patients with: adequate nutritional status, MNA ≥ 24; at risk for malnutrition, MNA between 17 and 23.5. proteincalorie undernutrition, MNA<17. This scale has been widely used, especially established as one of the most valid and most frequently used nutritional screening tools in older persons (Kaiser et al., 2010; Vellas et al., 1999).
Changes in Balance | The outcomes will be assessed at 5 time points: day before hospital discharge post-operation(Day 0), around 6±2 weeks post operation, around 3-month, 6-month and 12-month post operation.
  The 14-item Berg Balance Scale (BBS) will be used to measure elderly people's balance (Berg, Wood-Dauphine, Williams, & Gayton, 1989). It is an easily administrated tool and quick assessment in 10-15 minutes. Each item was scored from 0 (not at all) to 4 (all the time) with the sum score ranged from 0-56. The higher scores indicate better balance function and the score bellowing 45 points indicates the elderly is at fall risk. The BBS has been translated into Chinese and showed satisfying reliability and validity (Lima, Ricci, Nogueira, & Perracini, 2018).
Changes in Muscle strength and Endurance in Upper Limbs | The outcomes will be assessed at 5 time points: day before hospital discharge post-operation(Day 0), around 6±2 weeks post operation, around 3-month, 6-month and 12-month post operation.
  We will use Jamar grip strength meter to measure the strength of right and left upper limbs. Grip strength meter provided good reliability and validity for measuring muscle strength in the past studies (Cuesta-Vargas & Hilgenkamp, 2015; Silva et al., 2019). Patients will be asked to stand up, put arms by sides, and hold the meter to make a fist with maximal force for two times to record upper limbs strength.
Changes in Muscle strength and Endurance in Lower Limbs | The outcomes will be assessed at 5 time points: day before hospital discharge post-operation(Day 0), around 6±2 weeks post operation, around 3-month, 6-month and 12-month post operation.
  We will use microFET 2 to measure the strength of right and left hip flexor muscle. MicroFET 2 provided good reliability and validity for measuring muscle strength in the past studies (Cuesta-Vargas & Hilgenkamp, 2015; Silva et al., 2019). Patients will be seated on the chair. The researcher will put the microFET 2 on the upper edge of knee, and then let patient maintain the thigh raise for four seconds to record the strength of right and left hip flexor muscle.
Changes in Functional Mobility | The outcomes will be assessed at 5 time points: day before hospital discharge post-operation(Day 0), around 6±2 weeks post operation, around 3-month, 6-month and 12-month post operation.
  The Timed Up and Go test (TUG) is a frequently used clinical performance-based evaluation of a person's mobility, balance, walking ability, and fall risk (Herman et al., 2011). The patient gets up from an armchair, goes three meters, turns around, walks back, and then sits down again while being watched and timed (Podsiadlo & Richardson, 1991). A person who needs more than 12 seconds to finish the TUG runs the danger of falling. (Lusardi et al., 2017). The test is a reliable and valid test for quantifying functional mobility and is easily included as part of the medical examination.

CONTACTS AND LOCATIONS:
Overall Officials: Yeur-Hur Lai, Professor, Study Chair — School of Nursing, College of Medicine, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Chie WC, Yang CH, Hsu C, Yang PC. Quality of life of lung cancer patients: validation of the Taiwan Chinese version of the EORTC QLQ-C30 and QLQ-LC13. Qual Life Res. 2004 Feb;13(1):257-62. doi: 10.1023/B:QURE.0000015295.74812.06. PMID 15058806
- [Background] Kroenke K, Spitzer RL, Williams JB, Monahan PO, Lowe B. Anxiety disorders in primary care: prevalence, impairment, comorbidity, and detection. Ann Intern Med. 2007 Mar 6;146(5):317-25. doi: 10.7326/0003-4819-146-5-200703060-00004. PMID 17339617
- [Background] Remes O, Brayne C, van der Linde R, Lafortune L. A systematic review of reviews on the prevalence of anxiety disorders in adult populations. Brain Behav. 2016 Jun 5;6(7):e00497. doi: 10.1002/brb3.497. eCollection 2016 Jul. PMID 27458547
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Hinz A, Klein AM, Brahler E, Glaesmer H, Luck T, Riedel-Heller SG, Wirkner K, Hilbert A. Psychometric evaluation of the Generalized Anxiety Disorder Screener GAD-7, based on a large German general population sample. J Affect Disord. 2017 Mar 1;210:338-344. doi: 10.1016/j.jad.2016.12.012. Epub 2016 Dec 18. PMID 28088111
- [Background] Lowe B, Decker O, Muller S, Brahler E, Schellberg D, Herzog W, Herzberg PY. Validation and standardization of the Generalized Anxiety Disorder Screener (GAD-7) in the general population. Med Care. 2008 Mar;46(3):266-74. doi: 10.1097/MLR.0b013e318160d093. PMID 18388841
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Accuracy of Patient Health Questionnaire-9 (PHQ-9) for screening to detect major depression: individual participant data meta-analysis. BMJ. 2019 Apr 12;365:l1781. doi: 10.1136/bmj.l1781. No abstract available. PMID 30979729
- [Background] Lee YH, Hu CC, Humphris G, Huang IC, You KL, Jhang SY, Chen JS, Lai YH. Screening for fear of cancer recurrence: Instrument validation and current status in early stage lung cancer patients. J Formos Med Assoc. 2020 Jun;119(6):1101-1108. doi: 10.1016/j.jfma.2019.10.007. Epub 2019 Oct 31. PMID 31677865
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] He Y, Meng Z, Jia Q, Hu F, He X, Tan J, Zhang G, Li X, Zhang J, Zhang Q, Liu L, Zhao L, Li J, Wang Y, Qian Y, Hou S, Liu H, Wang S, Wang R, Zheng W, Hu T, Liu N, Upadhyaya A, Liu Y. Sleep Quality of Patients with Differentiated Thyroid Cancer. PLoS One. 2015 Jun 17;10(6):e0130634. doi: 10.1371/journal.pone.0130634. eCollection 2015. PMID 26083787
- [Background] Van Onselen C, Dunn LB, Lee K, Dodd M, Koetters T, West C, Paul SM, Aouizerat BE, Wara W, Swift P, Miaskowski C. Relationship between mood disturbance and sleep quality in oncology outpatients at the initiation of radiation therapy. Eur J Oncol Nurs. 2010 Dec;14(5):373-9. doi: 10.1016/j.ejon.2009.12.002. Epub 2010 Jan 18. PMID 20080444
- [Background] Tsai PS, Wang SY, Wang MY, Su CT, Yang TT, Huang CJ, Fang SC. Psychometric evaluation of the Chinese version of the Pittsburgh Sleep Quality Index (CPSQI) in primary insomnia and control subjects. Qual Life Res. 2005 Oct;14(8):1943-52. doi: 10.1007/s11136-005-4346-x. PMID 16155782
- [Background] Godin, G. The Godin-Shephard Leisure-Time Physical Activity Questionnaire. Health Fit J Can. 2011; 4: 18-22.
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Kaiser MJ, Bauer JM, Ramsch C, Uter W, Guigoz Y, Cederholm T, Thomas DR, Anthony PS, Charlton KE, Maggio M, Tsai AC, Vellas B, Sieber CC; Mini Nutritional Assessment International Group. Frequency of malnutrition in older adults: a multinational perspective using the mini nutritional assessment. J Am Geriatr Soc. 2010 Sep;58(9):1734-8. doi: 10.1111/j.1532-5415.2010.03016.x. PMID 20863332
- [Background] Vellas B, Guigoz Y, Garry PJ, Nourhashemi F, Bennahum D, Lauque S, Albarede JL. The Mini Nutritional Assessment (MNA) and its use in grading the nutritional state of elderly patients. Nutrition. 1999 Feb;15(2):116-22. doi: 10.1016/s0899-9007(98)00171-3. PMID 9990575
- [Background] Berg KO, Wood-Dauphinee SL, Williams JI, Gayton D. Measuring balance in the elderly: preliminary development of an instrument. Physiother Can. 1989; 41(6):304-11.
- [Background] Lima CA, Ricci NA, Nogueira EC, Perracini MR. The Berg Balance Scale as a clinical screening tool to predict fall risk in older adults: a systematic review. Physiotherapy. 2018 Dec;104(4):383-394. doi: 10.1016/j.physio.2018.02.002. Epub 2018 Feb 15. PMID 29945726
- [Background] Cuesta-Vargas A, Hilgenkamp T. Reference Values of Grip Strength Measured with a Jamar Dynamometer in 1526 Adults with Intellectual Disabilities and Compared to Adults without Intellectual Disability. PLoS One. 2015 Jun 8;10(6):e0129585. doi: 10.1371/journal.pone.0129585. eCollection 2015. PMID 26053852
- [Background] Herman T, Giladi N, Hausdorff JM. Properties of the 'timed up and go' test: more than meets the eye. Gerontology. 2011;57(3):203-10. doi: 10.1159/000314963. Epub 2010 May 20. PMID 20484884
- [Background] Lusardi MM, Fritz S, Middleton A, Allison L, Wingood M, Phillips E, Criss M, Verma S, Osborne J, Chui KK. Determining Risk of Falls in Community Dwelling Older Adults: A Systematic Review and Meta-analysis Using Posttest Probability. J Geriatr Phys Ther. 2017 Jan/Mar;40(1):1-36. doi: 10.1519/JPT.0000000000000099. PMID 27537070
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946